CLINICAL TRIAL: NCT00681096
Title: Causes of Low Back Pain in Nurses in Israeli Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Osnat Aharon, RN, MA, Hillel Yaffe Medical Center, Orthopedics Dept. A
Other Study IDs: 25/2008
Record Dates: First submitted 2008-05-18; First posted 2008-05-21 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Low Back Pain
Keywords: Low back pain in nurses
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
An examination of the various factors that cause lower back pain in nurses in four hospitals in Israel such as; socio-demographic, professional, posture while ambulating patients and job environment.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in orthopedics, surgical, intensive care and internal medicine units

Exclusion Criteria:

* All others

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses working in 4 Israeli hospitals
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2008-06

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel